CLINICAL TRIAL: NCT04088942
Title: A Randomized Open-label, Superiority, Multicenter, Two-arm Intervention Study of the Effect of "High-intensity" vs. 'Low-intensity' Smoking Cessation Intervention in Active Smokers With COPD
Brief Title: TOBacco STOP in Chronic Obstructive Pulmonary Disease-Trial - Study Protocol
Acronym: TOB-STOP-COP
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No funding
Sponsor: Pradeesh Sivapalan (Other)
Responsible Party: Sponsor-Investigator, Pradeesh Sivapalan, MD, PhD student, Chronic Obstructive Pulmonary Disease Trial Network, Denmark
Organization: Chronic Obstructive Pulmonary Disease Trial Network, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Protocol_TOB-STOP-COP_MISJUJ
Record Dates: First submitted 2019-09-11; First posted 2019-09-13 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; Smoking Cessation; Lung Diseases, Obstructive; Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease; Randomized Controlled Trial; Smoking Cessation; Behavioural support; varenicline; exacerbations
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking Cessation; Lung Diseases, Obstructive

STUDY DESIGN:
Intervention Model Description: This study will be performed as a randomized, open label, superiority, 2-arm intervention study in active smokers with COPD. A total of 600 participants will be included with startup 1st January 2020 and is expected to be completed 3 years later, January 2023. Participants are randomized (random allocation) 1:1 to a "low-intensity group" and a "high-intensity group". Stratified for age (>65 years vs. ≤65 years) and number of daily cigarettes (>10/day vs. ≤10/day). Blocked randomization through REDCap with blocks of varying sizes (4-8), which will not be disclosed. Participants, their data and laboratory specimens etc. will be assigned a coded identification number (ID) to maintain participant confidentiality.
  Participants will be randomized to either a low-intensity or a high-intensity smoking cessation intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-intensity group (Experimental): Will receive "high-intensity" intervention, which is a combination of pharmacological (varenicline) and behavioural support, described later.
  Interventions: Other: High-intensity smoking cessation intervention
- Low-intensity group (Active Comparator): Encouraged to quit smoking via own doctor and is prescribed varenicline.
  Interventions: Drug: Low-intensity smoking cessation intervention

INTERVENTIONS:
Other: High-intensity smoking cessation intervention — 1. Varenicline for 12 weeks - Day 1-3: 0.5 mg daily. Dag 4-7: 0.5 mg two times daily. Thereafter 1 mg 2 times daily.
  2. Group-sessions in 6 months:
  Preparation phase: 5 sessions Day 1-14: 5 sessions Day 15-30: 5 sessions Day 31-60: 5 sessions Day 61-90: 5 sessions Day 90-180: 5 sessions c) Hotline and scheduled phone consultations:
  1. A hotline is established which the high-intensity group can call.
  2. Weekly calls to all patients in the project for 26 weeks. Call for 5-10 min. If the patient has not had relapse, there will be called week 34 and week 42. If the patient has had relapse, calls continue until relapse-free for 10 weeks, then week 34 and week 42.
     d) Buddy-arrangement: i. Patients who have completed the program and have become smoke-free, are matched with new ones in the program. A meeting frequency of approx. every 7-14 days. The first patients are matched with patients from pulmonary medical outpatient clinic who have ceased smoking.
  Arms: High-intensity group
Drug: Low-intensity smoking cessation intervention — Varenicline prescribed for 12 weeks - Day 1-3: 0.5 mg daily. Dag 4-7: 0.5 mg two times daily. Thereafter 1 mg 2 times daily.
  Arms: Low-intensity group

SUMMARY:
Background:

Cigarette smoking is the leading cause of chronic obstructive pulmonary disease (COPD) and it contributes to the development of many other serious diseases. Acute exacerbations of COPD (AECOPD) often lead to hospitalization. Severe hospitalization-requiring AECOPD carries very high economic costs for the healthcare system, and personal costs for patients. Smoking cessation in COPD for the healthcare system, and personal costs for patients. Smoking cessation in COPD patients is known to improve survival and reduce the number of AECOPD. However, smoking cessation interventions in these patients have only been successful for consistent smoking abstinence in 12 months in approximately 15-20%. Thus, more effective interventions are needed for this patient group.

Aims:

The aim of this study is to determine, among people with chronic obstructive pulmonary disease (COPD), whether a "high-intensive" smoking cessation intervention in comparison to a standard intervention can lead to permanent, >12 months, smoking cessation in a higher proportion.

Methods:

This study is a randomized trial in active smokers with COPD and who have lost less than 50% lung function. A total of 600 participants will be randomly assigned 1:1 to either a standard treatment (guideline-based municipal smoking cessation programme, "low intensity" group), or an intervention group ("high-intensity" group), which consists of group sessions, telephone consultations, behavior design, hotline, "buddy-matching" (smoker matched with COPD patient who stopped). Both groups will receive pharmacological smoking cessation.

Discussion:

The potential benefit of this project is to prevent smoking-related exacerbations of COPD and thereby reduce logistics and costs of hospitalization and treatment of COPD. In addition, the project can potentially benefit from increasing the quality of life and longevity of COPD patients and reducing the risk of developing lung cancer and other smoking-related diseases.

DETAILED DESCRIPTION:
Hypothesis:

A "high-intensity" smoking cessation intervention is superior in leading to permanent (>12 months) smoking cessation in active smokers with COPD than does a standard, guideline-based municipal smoking cessation intervention.

Secondary hypothesis: The progression of COPD will be reduced in the "high intensity group", and this will result in limited loss of lung function, a reduced number of exacerbations of COPD, improved mental health and self-rated health.

Rationale:

Smoking cessation in COPD patients improves survival and reduces the number of exacerbations. Unfortunately, relatively few COPD patients are successful in permanently stopping to smoke, even with pharmacological help.

Primary aim: to determine if a high-intensity intervention in comparison to a low-intensity intervention can lead to persistent (>12 months) anamnestic and biochemical smoking cessation in more active smokers with COPD.

Secondary aim 1: to investigate, within the randomized study design, long-term follow-up over 2 years and 5 years, whether the occurrence of depressive symptoms and anxiety symptoms is different in the "high-intensity" and "low-intensity" group. This is estimated by means of a. Depression questionnaires and b. Consumption of pharmaceuticals that are primarily prescribed for these conditions.

Secondary aim 2: to characterize changes in the respiratory microbiome between active smokers with COPD and COPD patients who have stopped smoking to find out whether the airway microbiome adapts/changes after smoking cessation.

Background:

COPD is a life-threatening and incurable lung disease characterized by persistent breathing problems and poor airflow in the lungs. Globally, it is estimated that approx. 250 million people have COPD and that approx. 3 million deaths annually, corresponding to 5% of all deaths worldwide, are caused by COPD. In Denmark, there are about 320,000 people with COPD, where approx. 5500 die due to COPD each year, making the disease the third most frequent cause of death in Denmark. Cigarette smoking is by far the most important cause of development of COPD by causing lung inflammation, which leads to release of oxidative radicals, and this in turn leads to destruction of lung tissue (both respiratory tissue and conductive tissue). Cigarette smokers have a higher incidence of respiratory symptoms and abnormal lung function, a greater annual decrease in FEV1 (forced expiratory volume for 1 second) and a greater mortality rate than non-smokers.

Acute exacerbations (worsening) of COPD (AECOPD) are associated with increased risk of mortality due to decreasing lung function and activity level and often lead to hospitalization. This is one of the biggest costs for the healthcare system for treatment of COPD. In addition, there is evidence that AECOPD increases the risk of myocardial infarction and strokes. In this way, smoking cessation will be the most effective intervention to stop the development of COPD, as well as increase survival and reduce morbidity. Overall, tobacco smoking thus increases mortality and serious morbidity as well as symptoms in COPD patients, and smoking cessation should be the top priority in treating COPD.

Current evidence of smoking cessation:

However, smoking cessation is only successful in a minority of patients with COPD. In an intervention study from 2011 (N = 499), after 12 months, only 18,6% of COPD patients treated with varenicline had still stopped smoking, while 5,6% of patients in the placebo group had obtained this. Despite a significant difference in absolute risk of 13% between the varenicline and placebo group, it is still >80% of COPD patients in the varenicline group who smoke after 12 months, which is not satisfactory.

In an observational study from 2008 among patients with COPD who participated in a new 1 year smoking cessation programme (N = 247), smoking cessation rates were as high as 52% after 1 year and 38% after 3 years. The results were compared with a group of COPD patients who received normal care (N = 231), in which smoking cessation rates were 7% after 1 year and 10% after 3 years. The smoking cessation program in the patients who participated in the new programme included a 2-week period of admission to hospitals, group sessions where nicotine replacement therapy (NRT) and exercise were recommended/advised in, and in addition telephone calls with specially trained staff who gave feedback and support for smoking cessation throughout the year. Although these results are very inspiring, the obvious weaknesses in the design leave open numerous possibilities for errors in the estimates. Such an advanced, multipoint smoking cessation has never been tested in a solid design like a randomized controlled trial.

Method:

Design:

Study A) A randomized open-label, superiority, multicenter, 2-arm intervention study, in which it is examined if a "high-intensity" intervention causes fewer people (diagnosed with COPD) to smoke after 12 months than in a "low-intensity" intervention in people diagnosed with COPD. The effect on survival for 12, 24 and 48 months, incidence of COPD exacerbations, number of admissions for all causes and cardiovascular admissions will also be analyzed at the same times.

Study B) Depression/anxiety within the framework of the randomized study ("high-intensity" vs. "low-intensity" group). Measured by means of questionnaires and by recording the prescription of drugs for depression and anxiety.

Study C) A microbiological study within the framework of the randomized study, which aims to investigate the respiratory microbiome and possibly changes in participants in the two randomized groups. Subgroup analyzes for participants who actively smoke vs. have ceased and exploratory analyzes to determine if the microbiome changes within 6 months after

Data collection:

The primary daily project management is handled by the project manager. In addition, a project group, consisting of health professionals from the departments involved, is trained to assist the project manager with recruitment, sampling and follow-up of participants. Recruitment in general practice is done by the project-trained nurse.

Upon entering the program and all visits in the future (after 1, 3, 6, 12, 24 and 36 months), the participant is summoned to a conversation with staff, asking if the participant smokes (yes vs. no), and if yes, how much. In addition, a urine sample is taken for cotinine analysis for biochemical verification of smoking status and standard blood samples to examine health status at these visits (analyzed on Department of Clinical Biochemistry, KBA). In addition, questionnaires: COPD Assessment Test (CAT), Medical Research Council dyspnea scale (MRC), and Hospital Anxiety and Depression Scale (HADS) are completed with the participant. In the case of inclusion and follow-up visits after 3, 6, 12, 24 and 36 months, spirometry is also carried out at regular intervals. Height measurement is done by inclusion in the study along with weight measurement, which is only further measured after 6, 12, 24 and 36 months to monitor BMI.

The Hamilton Depression scale (HAM-D) score is performed by inclusion, after 12, 24 and 36 months and if the score becomes high (≥25), i.e. that there is a high risk of developing depression, the participant is referred for examination for depression via their own doctor.

In addition, sputum samples are induced (with isotonic saline water) for microbiome analysis by inclusion of the study, and again after 12 months in the first 50 participants in the "high-intensity" group who quit smoking, and in the first 50 participants in the "low-intensity" group, who do not quit smoking.

Intervention:

600 active smokers with COPD will be included. Stratified for age (>65 years vs. 65 years) and number of daily cigarettes (>5/day vs. ≤5/day). There are randomized blocks of varying sizes (4-8). Block sizes will be concealed to investigators.

Participants will be randomized to one of the following two treatment groups:

1. "Low-intensity group": encouraged to quit smoking via own doctor and varenicline is prescribed for 12 weeks.
2. "High-intensity group": a. Varenicline for 12 weeks b. Group-sessions - in all 30 sessions divided into 6 months i. Preparation phase: 5 sessions ii. Day 1-14: 5 sessions iii. Day 15-30: 5 sessions iv. Day 31-60: 5 sessions v. Day 61-90: 5 sessions vi. Day 90-180: 5 sessions

Group sessions are controlled by:

I. Pulmonary Nurse [Mapping of different smoking patterns and different reasons for smoking. When is smoking the greatest? When in the process, smoking starts to fall. Dangerous situations regarding smoking relapses. Initial focus on nicotine-craving and coping methods] II. Pulmonary doctor [Lung function, Lung age, Anatomy, Physiology, Pathophysiology of lung cancer and COPD]. Focus on why smoking cessation is good. Is there anything you want to experience in your life that smoking can prevent? Either by death or because illness would prevent it? III. Psychologist [Focus on behavior before smoking and how this behavior is slowed down at an early stage. Coping by smoking. Cognitive smoking cessation strategies. Handle digito-oral habit].

IV. Physiotherapist [Training on how to improve general physical form. Forming individual training programs].

V. Dietician (focus on keeping weight (both ways), nutrition). Suggestions for what to eat by smoking craving.

c) Relationships and retention via these: i. Hotline and scheduled phone consultations:

1. A hotline is established which the "high-intensity group" can call.
2. Weekly calls to all participants in the project for 26 weeks. Call for 5-10 min. If the participant has not had relapse, there will be called week 34 and week 42. If the participant has had relapse, calls continue until relapse-free for 10 weeks, then week 34 and week 42.

   d) "Buddy-arrangement": i. Participants who have completed the program and have become smoke-free, are matched with new ones in the program. A meeting frequency of approx. every 7-14 days. The first participants are matched with patients from respiratory medicine outpatient clinic who have ceased smoking.

   Patients with COPD fear acute exacerbations since this increases dyspnea, cough, sputum and is associated with significant morbidity and mortality. Smoking cessation is the best intervention for exacerbations and progression of COPD in active smokers with COPD. The potential benefit of this project is to prevent smoking-related exacerbations of COPD and thereby reduce logistics and costs of hospitalization and treatment of COPD. In addition, the participants can potentially benefit from fewer mental depressions, increased self-rated quality of life and longevity of COPD patients and can reduce the risk of developing lung cancer (the leading cause of death in COPD patients with >50% lung function (FEV1) preserved) and other smoking-related diseases. Possibly, the project may also cause "healthy" smokers to stop smoking. Based on this, the investigators believe that the experiment is scientifically sound and that the trial participants will not be exposed to irresponsible risks.

ELIGIBILITY:
Inclusion Criteria:

* Competent and mature
* Have diagnosed COPD [spirometry verified and evaluated by pulmonary specialist]
* Current daily smoker [Minimum 1 cigarette daily]
* Have smoked minimum 20 pack years (1 pack year = 20 cigarettes daily in 1 year)
* Want to or try to stop smoking
* Do not mind taking varenicline or NRT during the trial
* Are willing to give blood and urine samples according to the protocol

Exclusion Criteria:

* Previously included in the trial
* Hospitalized with COPD-exacerbation within the last 24 months
* Are associated with hospital outpatient clinic for COPD disease treatment
* Have FEV1<50%.
* Pregnancy/breastfeeding
* Life expectancy less than 1 year
* Severe linguistic problems or inability to give informed consent
* Severe mental illness that is not controlled with medication
* Active alcohol or substance abuse
* Active cancer disease* *The person can participate if he or she has had a cancer disease that is now referred to as curative/radically treated. Basal cell carcinoma of the skin does not count as an exclusion criterion.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Anamnestic and biochemical* validated smoking cessation | 12 months after inclusion
  *Cotinine is analyzed in a urine sample, as validated point-prevalence for the last 7 days

SECONDARY OUTCOMES:
Number of admissions for exacerbations of COPD or death | Within 12 months after inclusion
Number of admissions for all causes or death | Within 12 months after inclusion
Number of cardiovascular events | Within 12 months after inclusion
  Defined as cardiovascular death, acute myocardial infarction or unstable angina pectoris
Changes in CAT-score (COPD Assessment Test) | 12 months after inclusion
  Range of CAT scores from 0-40. Higher scores denote a more severe impact of COPD on a patient's life.
Changes in FEV1 from baseline | 12 months after inclusion
Changes in BMI | 12 months after inclusion
  BMI loss more than 1 unit
Clinically relevant changes in HADS-score (Hospital Anxiety and Depression Scale) | 12 months after inclusion
  Each item on the questionnaire is scored from 0-3. A person can score between 0 and 21 for either anxiety or depression. Higher scores indicate a more greater risk of either anxiety or depression.
Occurrence of DNA from the following: M. catarrhalis, H. influenzae and P. aeruginosa | 12 months after inclusion
  These end-points are only examined on the first 50 who stop smoking from the "high-intensity" group against the first 50 who do not stop smoking from the "low-intensity" group.
Changes in the total lung microbiome | 12 months after inclusion
  These end-points are only examined on the first 50 who stop smoking from the "high-intensity" group against the first 50 who do not stop smoking from the "low-intensity" group.
Occurrence of smoking-related cancer | Within 12 months after inclusion
  Lung cancer, urothelial cancer, pancreatic cancer, esophageal cancer, pharyngeal cancer, laryngeal cancer, tongue cancer, oral cancer, tonsil cancer
Number of admissions requiring non-invasive ventilation (NIV) treatment or admissions to intensive care or death | Within 12 months after inclusion
Changes in status from MRC-dyspnea score from < 3 to 3 ≥ (Medical Research Council dyspnea scale) | 12 months after inclusion
  The scale ranges from 1-5, higher score indicate a greater extent to which patients' breathlessness affects their mobility. Patients who score 3, 4 or 5 on MRC-dyspnea scale may be offered rehabilitation according to international recommendations.

OTHER OUTCOMES:
Occurrence of depression | Within 36 months after inclusion
  1. Admission to psychiatry with depression as primary diagnosis
  2. New start of antidepressant treatment after baseline
  3. Clinically relevant changes in HADS score over 36 months
  4. Changes in status from HAM-D score from baseline over 36 months
Number of days during antidepressant treatment | 36 months after inclusion
Changes in FEV1 | 36 months after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Jens-Ulrik S Jensen, MD, PhD, Principal Investigator — Herlev-Gentofte Hospital, COP:TRIN
Locations (4):
- Denmark (4):
  - Bispebjerg University Hospital, Copenhagen
  - Hvidovre University Hospital, Copenhagen
  - North Zealand Hospital, Copenhagen
  - Department of Internal medicine, Herlev & Gentofte Universtity Hospital, Hellerup

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] "Global Strategy for the Diagnosis, Management, and Prevention of Chronic Obstructive Lung Disease 2017 Report: GOLD Executive Summary." Claus F. Vogelmeier, Gerard J. Criner, Fernando J. Martinez, Antonio Anzueto, Peter J. Barnes, Jean Bourbeau, Bartolome R. Celli, Rongchang Chen, Marc Decramer, Leonardo M. Fabbri, Peter Frith, David M.G. Halpin, M. Victorina Lopez Varela, Masaharu Nishimura, Nicolas Roche, Roberto Rodriguez-Roisin, Don D. Sin, Dave Singh, Robert Stockley, Jorgen Vestbo, Jadwiga A. Wedzicha and Alvar Agusti. Eur Respir J 2017; 49: 1700214. Eur Respir J. 2017 Jun 22;49(6):1750214. doi: 10.1183/13993003.50214-2017. Print 2017 Jun. No abstract available. PMID 28642306
- [Background] Lopez-Campos JL, Tan W, Soriano JB. Global burden of COPD. Respirology. 2016 Jan;21(1):14-23. doi: 10.1111/resp.12660. Epub 2015 Oct 23. PMID 26494423
- [Background] Tonnesen P. Smoking cessation and COPD. Eur Respir Rev. 2013 Mar 1;22(127):37-43. doi: 10.1183/09059180.00007212. PMID 23457163
- [Background] Maurer J, Rebbapragada V, Borson S, Goldstein R, Kunik ME, Yohannes AM, Hanania NA; ACCP Workshop Panel on Anxiety and Depression in COPD. Anxiety and depression in COPD: current understanding, unanswered questions, and research needs. Chest. 2008 Oct;134(4 Suppl):43S-56S. doi: 10.1378/chest.08-0342. PMID 18842932
- [Background] Mammen MJ, Sethi S. COPD and the microbiome. Respirology. 2016 May;21(4):590-9. doi: 10.1111/resp.12732. Epub 2016 Jan 27. PMID 26852737
- [Background] Paggiaro PL, Chanez P, Holz O, Ind PW, Djukanovic R, Maestrelli P, Sterk PJ. Sputum induction. Eur Respir J Suppl. 2002 Sep;37:3s-8s. doi: 10.1183/09031936.02.00000302. No abstract available. PMID 12361361
- [Background] Jespersen CM, Als-Nielsen B, Damgaard M, Hansen JF, Hansen S, Helo OH, Hildebrandt P, Hilden J, Jensen GB, Kastrup J, Kolmos HJ, Kjoller E, Lind I, Nielsen H, Petersen L, Gluud C; CLARICOR Trial Group. Randomised placebo controlled multicentre trial to assess short term clarithromycin for patients with stable coronary heart disease: CLARICOR trial. BMJ. 2006 Jan 7;332(7532):22-7. doi: 10.1136/bmj.38666.653600.55. Epub 2005 Dec 8. PMID 16339220
- [Result] Hersh CP, DeMeo DL, Al-Ansari E, Carey VJ, Reilly JJ, Ginns LC, Silverman EK. Predictors of survival in severe, early onset COPD. Chest. 2004 Nov;126(5):1443-51. doi: 10.1378/chest.126.5.1443. PMID 15539711
- [Result] Au DH, Bryson CL, Chien JW, Sun H, Udris EM, Evans LE, Bradley KA. The effects of smoking cessation on the risk of chronic obstructive pulmonary disease exacerbations. J Gen Intern Med. 2009 Apr;24(4):457-63. doi: 10.1007/s11606-009-0907-y. Epub 2009 Feb 5. PMID 19194768
- [Result] Tashkin D, Kanner R, Bailey W, Buist S, Anderson P, Nides M, Gonzales D, Dozier G, Patel MK, Jamerson B. Smoking cessation in patients with chronic obstructive pulmonary disease: a double-blind, placebo-controlled, randomised trial. Lancet. 2001 May 19;357(9268):1571-5. doi: 10.1016/s0140-6736(00)04724-3. PMID 11377644
- [Result] Alberg AJ, Brock MV, Ford JG, Samet JM, Spivack SD. Epidemiology of lung cancer: Diagnosis and management of lung cancer, 3rd ed: American College of Chest Physicians evidence-based clinical practice guidelines. Chest. 2013 May;143(5 Suppl):e1S-e29S. doi: 10.1378/chest.12-2345. PMID 23649439
- [Result] Wang Q, Bourbeau J. Outcomes and health-related quality of life following hospitalization for an acute exacerbation of COPD. Respirology. 2005 Jun;10(3):334-40. doi: 10.1111/j.1440-1843.2005.00718.x. PMID 15955146
- [Result] Hurst JR, Vestbo J, Anzueto A, Locantore N, Mullerova H, Tal-Singer R, Miller B, Lomas DA, Agusti A, Macnee W, Calverley P, Rennard S, Wouters EF, Wedzicha JA; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints (ECLIPSE) Investigators. Susceptibility to exacerbation in chronic obstructive pulmonary disease. N Engl J Med. 2010 Sep 16;363(12):1128-38. doi: 10.1056/NEJMoa0909883. PMID 20843247
- [Result] Rothnie KJ, Yan R, Smeeth L, Quint JK. Risk of myocardial infarction (MI) and death following MI in people with chronic obstructive pulmonary disease (COPD): a systematic review and meta-analysis. BMJ Open. 2015 Sep 11;5(9):e007824. doi: 10.1136/bmjopen-2015-007824. PMID 26362660
- [Result] Portegies ML, Lahousse L, Joos GF, Hofman A, Koudstaal PJ, Stricker BH, Brusselle GG, Ikram MA. Chronic Obstructive Pulmonary Disease and the Risk of Stroke. The Rotterdam Study. Am J Respir Crit Care Med. 2016 Feb 1;193(3):251-8. doi: 10.1164/rccm.201505-0962OC. PMID 26414484
- [Result] Tashkin DP, Rennard S, Taylor Hays J, Lawrence D, Marton JP, Lee TC. Lung function and respiratory symptoms in a 1-year randomized smoking cessation trial of varenicline in COPD patients. Respir Med. 2011 Nov;105(11):1682-90. doi: 10.1016/j.rmed.2011.04.016. Epub 2011 May 31. PMID 21621992
- [Result] Tonnesen P, Mikkelsen K, Bremann L. Nurse-conducted smoking cessation in patients with COPD using nicotine sublingual tablets and behavioral support. Chest. 2006 Aug;130(2):334-42. doi: 10.1378/chest.130.2.334. PMID 16899830
- [Result] Hartmann-Boyce J, Hong B, Livingstone-Banks J, Wheat H, Fanshawe TR. Additional behavioural support as an adjunct to pharmacotherapy for smoking cessation. Cochrane Database Syst Rev. 2019 Jun 5;6(6):CD009670. doi: 10.1002/14651858.CD009670.pub4. PMID 31166007
- [Result] Strassmann R, Bausch B, Spaar A, Kleijnen J, Braendli O, Puhan MA. Smoking cessation interventions in COPD: a network meta-analysis of randomised trials. Eur Respir J. 2009 Sep;34(3):634-40. doi: 10.1183/09031936.00167708. Epub 2009 Apr 8. PMID 19357145
- [Result] van Eerd EA, van der Meer RM, van Schayck OC, Kotz D. Smoking cessation for people with chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2016 Aug 20;2016(8):CD010744. doi: 10.1002/14651858.CD010744.pub2. PMID 27545342
- [Result] Rosen LJ, Galili T, Kott J, Goodman M, Freedman LS. Diminishing benefit of smoking cessation medications during the first year: a meta-analysis of randomized controlled trials. Addiction. 2018 May;113(5):805-816. doi: 10.1111/add.14134. Epub 2018 Jan 29. PMID 29377409
- [Result] Sundblad BM, Larsson K, Nathell L. High rate of smoking abstinence in COPD patients: Smoking cessation by hospitalization. Nicotine Tob Res. 2008 May;10(5):883-90. doi: 10.1080/14622200802023890. PMID 18569763
- [Result] Schneider C, Jick SS, Bothner U, Meier CR. COPD and the risk of depression. Chest. 2010 Feb;137(2):341-7. doi: 10.1378/chest.09-0614. Epub 2009 Oct 3. PMID 19801582
- [Result] Eisner MD, Blanc PD, Yelin EH, Katz PP, Sanchez G, Iribarren C, Omachi TA. Influence of anxiety on health outcomes in COPD. Thorax. 2010 Mar;65(3):229-34. doi: 10.1136/thx.2009.126201. PMID 20335292
- [Result] Pooler A, Beech R. Examining the relationship between anxiety and depression and exacerbations of COPD which result in hospital admission: a systematic review. Int J Chron Obstruct Pulmon Dis. 2014 Mar 29;9:315-30. doi: 10.2147/COPD.S53255. eCollection 2014. PMID 24729698
- [Result] Yohannes AM, Alexopoulos GS. Depression and anxiety in patients with COPD. Eur Respir Rev. 2014 Sep;23(133):345-9. doi: 10.1183/09059180.00007813. PMID 25176970
- [Result] Taylor G, McNeill A, Girling A, Farley A, Lindson-Hawley N, Aveyard P. Change in mental health after smoking cessation: systematic review and meta-analysis. BMJ. 2014 Feb 13;348:g1151. doi: 10.1136/bmj.g1151. PMID 24524926
- [Result] Dy R, Sethi S. The lung microbiome and exacerbations of COPD. Curr Opin Pulm Med. 2016 May;22(3):196-202. doi: 10.1097/MCP.0000000000000268. PMID 26964078
- [Result] Garcia-Nunez M, Millares L, Pomares X, Ferrari R, Perez-Brocal V, Gallego M, Espasa M, Moya A, Monso E. Severity-related changes of bronchial microbiome in chronic obstructive pulmonary disease. J Clin Microbiol. 2014 Dec;52(12):4217-23. doi: 10.1128/JCM.01967-14. Epub 2014 Sep 24. PMID 25253795
- [Derived] Hartmann-Boyce J, Theodoulou A, Farley A, Hajek P, Lycett D, Jones LL, Kudlek L, Heath L, Hajizadeh A, Schenkels M, Aveyard P. Interventions for preventing weight gain after smoking cessation. Cochrane Database Syst Rev. 2021 Oct 6;10(10):CD006219. doi: 10.1002/14651858.CD006219.pub4. PMID 34611902
- [Derived] Saeed MI, Sivapalan P, Eklof J, Ulrik CS, Pisinger C, Lapperre T, Tonnesen P, Hoyer N, Janner J, Karlsson ML, Bech CS, Marsa K, Godtfredsen N, Brondum E, Munk B, Raaschou M, Browatzski A, Lutken P, Jensen JS. TOB-STOP-COP (TOBacco STOP in COPd trial): study protocol-a randomized open-label, superiority, multicenter, two-arm intervention study of the effect of "high-intensity" vs. "low-intensity" smoking cessation intervention in active smokers with chronic obstructive pulmonary disease. Trials. 2020 Aug 21;21(1):730. doi: 10.1186/s13063-020-04653-z. PMID 32825845
- See also: World Health Organization. Chronic obstructive pulmonary disease fact sheet. — http://www.who.int/en/news-room/fact-sheets/detail/chronic-obstructive-pulmonary-disease-(copd)
- See also: Danish Lung Association and www.lunge.dk. Key numbers on pulmonary diseases — https://www.lunge.dk/lunger/viden-noegletal-om-lungesygdomme